CLINICAL TRIAL: NCT06319456
Title: A Global Multicenter, Open Label, Randomized Phase III Confirmatory Study of Lisaftoclax (APG-2575) in Combination With Acalabrutinib Versus Immunochemotherapy in Patients With Newly Diagnosed Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (GLORA-2).
Brief Title: A Global Study of Lisaftoclax (APG-2575) Combined With Acalabrutinib Versus Immunochemotherapy for Newly Diagnosed CLL/SLL.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ascentage Pharma Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APG2575CC301
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: CLL/SLL
Keywords: CLL/SLL; Lisaftoclax; APG-2575
MeSH Terms: interventions — Lisaftoclax; acalabrutinib; fludarabine; Rituximab; Chlorambucil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lisaftoclax (APG-2575) combined with Acalabrutinib (Experimental)
  Interventions: Drug: Lisaftoclax (APG-2575); Drug: Acalabrutinib
- Immunochemotherapy regimens (Active Comparator)
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide，CTX; Drug: Rituximab; Drug: Chlorambucil

INTERVENTIONS:
Drug: Lisaftoclax (APG-2575) — QD, oral administration, every 28 days for a dosing cycle.
  Arms: Lisaftoclax (APG-2575) combined with Acalabrutinib
Drug: Acalabrutinib — BID, oral administration, every 28 days for a dosing cycle.
  Arms: Lisaftoclax (APG-2575) combined with Acalabrutinib
Drug: Fludarabine — Every 28 days for a treatment cycle, administration of 6 cycles.
  Arms: Immunochemotherapy regimens
Drug: Cyclophosphamide，CTX — Every 28 days for a treatment cycle, administration of 6 cycles.
  Arms: Immunochemotherapy regimens
Drug: Rituximab — Every 28 days for a treatment cycle, administration of 6 cycles.
  Arms: Immunochemotherapy regimens
Drug: Chlorambucil — Every 28 days for a treatment cycle, administration of 6 cycles.
  Arms: Immunochemotherapy regimens

SUMMARY:
This is a global, multicenter, randomized, open-label, Phase III confirmatory study to investigate the efficacy and safety of Lisaftoclax (APG-2575) in combination with Acalabrutinib in patients with newly diagnosed CLL/SLL.

DETAILED DESCRIPTION:
The patients with newly diagnosed CLL/SLL, who have met all required eligibility criteria, will be randomized to the investigational group (Lisaftoclax in combination with Acalabrutinib) or the control group (immunochemotherapy, CIT).

ELIGIBILITY:
1. CLL/SLL must be diagnosed according to the IWCLL NCI-WG Guidelines (2018 edition) and meet at least one of the criteria requiring treatment.
2. With a measurable disease.
3. ECOG score 0-2.
4. QTcF interval: ≤450ms in males, ≤470ms in females.
5. Adequate bone marrow function independent of growth factor support.
6. Adequate liver, kidney and coagulation function.
7. Males and females of childbearing potential, and their partners voluntarily use effective contraceptive measures throughout the treatment and for at least three months after the last dose of the study drug. Male patients must avoid donation from the first dose of the study drug to three months after the last dose of the study drug.
8. Female patients of childbearing potential have negative serum pregnancy test results within 14 days prior to the first dose of the study drug.
9. Patients must be able to understand and voluntarily sign an informed consent form approved by the Ethics Committee (EC) before commencing any screening or study specific procedures.
10. Must be willing and able to complete research procedures and follow-up examinations.

Exclusion Criteria:

1. Any previous CLL specific treatment.
2. Failure to fully recover adequately from prior surgical procedures at the discretion of the investigator. Patients who receive a major surgery within 28 days prior to the first dose of the study drug or who receive a minor surgery (excluding biopsy) within 14 days prior to the initiation of the study.
3. Presence of significant cardiovascular disease within 6 months prior to study entry.
4. A history of significant kidney, neurological, psychiatric, pulmonary, endocrine, metabolic, immune, cardiovascular, or liver disease, which will have an adverse effect on the patient if he/she participates in the study, at the discretion of the investigator.
5. Patients who require warfarin or other anticoagulants or active hemorrhage occur within 2 months before study entry.
6. Known to have hypersensitivity to the drug ingredient or its analogues.
7. Pregnant or lactating female patients and patients who are expected to become pregnant during the study period or within 3 months after the last dose.
8. Patients who have history of other active malignant tumor other than CLL/SLL within 3 years before study entry.
9. With a malabsorption syndrome or other conditions unsuitable for enteral administration.
10. Other clinically significant uncontrolled symptoms.
11. With primary active autoimmune disease and connective tissue disease.
12. Any other circumstances or conditions that would, at the discretion of the investigator, make the patient unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Estimated)
Dates: Start 2024-04-07 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Progress Free Survival (PFS) | Up to 1 year
  PFS is defined as the time from randomization to disease progression(PD) or death from any cause.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 1 year
  ORR is defined as the proportion of patients who have achieved CR, CRi or PR.
Minimal Residual Disease (MRD) negativity rate | Up to 1 year
  To observe the proportion of patients with MRD negativity in bone marrow, peripheral blood, either or both.
Safety evaluation based on the adverse event concurrence | Up to 1 year
  Number of treatment emergent adverse events (TEAEs) and treatment related adverse events (TRAEs) will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Lugui Qiu, M.D., Ph.D., Principal Investigator — Hematology Hospital of the Chinese Academy of Medical Sciences; Keshu Zhou, M.D., Ph.D., Principal Investigator — Henan Province Cancer Hospital
Locations (6):
- China (6):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Henan Provincial Cancer Hospital, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hematology Hospital of the Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality